CLINICAL TRIAL: NCT04455607
Title: The Influence of a Perturbation Training on Balance Recovery of Old Adults - a Randomized Controlled Trial
Brief Title: Perturbation Training to Improve Balance Recovery of Old Adults
Acronym: BalancING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Sor 396-16 CTIL
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2020-10

CONDITIONS: Old Adults

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Random perturbation training
  Interventions: Behavioral: perturbation training
- control group (Active Comparator): Block perturbation training
  Interventions: Behavioral: perturbation training

INTERVENTIONS:
Behavioral: perturbation training — A Randomized control trial we will compare two perturbation motor learning paradigms with different challenge level of the practice condition (i.e. blocked practice vs random practice). According to motor learning theory we hypothesize that a) healthy older adults will benefit more from random practice. The purpose of this stage is to investigate the effects of task practice order (random vs blocked) on motor learning (i.e. responding to perturbations during walking) in older adults. According to motor learning theory we hypothesize that a) healthy older adults will benefit more from the random motor learning approach as compared to using blocked practice.

SUMMARY:
Falls are major contributors for immobility and independency. Most falls in older adults occur during walking after a sudden unexpected loss of balance. It was well-established that balance can be improved by performance of a training program that provides perturbation (unexpected perturbations of balance). The main aim of the current study is to investigate the effects of two perturbation-training methods: 1) random perturbation training; vs. 2) block (non-random) perturbation training. We also aim to explore brain area's (as measured by MRI) that are related to balance function in older adults.

We hypothesize that response to an unexpected loss of balance is the balance responses will be improved in both training methods, but more in the random training method. We also hypothesize that brain function as seen in MRI will be improved in both training methods, more in the random training method.

As far as we know, there is a lack of studies investigating the learning effect of random vs. block non-random training on balance recovery responses while walking and exposure to unexpected loss of balance and on brain function.

DETAILED DESCRIPTION:
Goals:

1. Determine the relationship between gait stability (as measured in the Lab) and brain function (MRI) in 50 old (70 years old and over) and 10 young adults (20-40 years old) that represent heathy brain.
2. To determine which of the training intervention methods (25 older adults that participate in random training vs. 25 older adults that participate in block non-random training) are more beneficial for balance recovery responses and for improved brain function.

Methods: This study is a clinical investigation study. First stage - Individuals that show an interest in participating in the study will be exposed to a brief interview before further testing is performed to see if they fit the inclusion-exclusion criteria. Individuals who pass the interview a screening, and physical examination and the additional questionnaires and functional tests described below.

Second stage - Testing different motor learning paradigms for improving balance recovery ability: A convenience sample of 60 healthy subjects (10 young's, 50 older adults) will be recruited. After testing their clinical balance performance (Berg balance test, 6-minutes' walk and get up and go) and cognitive function (MOCA), All testing will occur on a specific motor-driven surface perturbation treadmill (BaMPer). The Gait protocol will include about 10-20 minutes of comfortable pace walking, than progressive unexpected surface perturbations will be added. The same protocol will be performed with during standing condition. Subjects will also walk on the treadmill without perturbations. The order of the different test conditions will be randomized.

Outcome measures: The stepping threshold as measured by the distance of the platform movements in centimeters will be measured. Quantitative parameters of the compensatory stepping/ and motor ability (i.e., step reaction time, step time, step length), descriptive parameters of the stepping strategy after perturbation

(i.e., arm responses, upper body responses, leg step threshold and fall threshold). In addition, we will be testing the correlation between brain activity and anatomy using brain imaging in 10 young and 50 older adults and correlate with balance/motor function.

The aims of this study are to determine the relationship between the different requirements for gait stability (walking without perturbations, ability to overcome small perturbations, ability to overcome larger perturbations and, largest recoverable perturbation during walking) and brain function and anatomy. The research hypothesis: there is a correlation between the age related atrophies in areas of the brain and functional capacity

Third stage - A Randomized control trial we will compare two perturbation motor learning paradigms with different challenge level of the practice condition (i.e. blocked practice vs random practice). According to motor learning theory we hypothesize that a) healthy older adults will benefit more from random practice. The purpose of this stage is to investigate the effects of task practice order (random vs blocked) on motor learning (i.e. responding to perturbations during walking) in older adults. According to motor learning theory we hypothesize that a) healthy older adults will benefit more from the random motor learning approach as compared to using blocked practice.

ELIGIBILITY:
Inclusion Criteria:

1. 70 years and older (with the young age of 20-40)
2. able to walk independently (without utilities treadmill or stick);
3. Be asked to invent a medical certificate which allows participation in exercise that requires walking twice a week.

Exclusion Criteria:

1. suffering from ischaemic heart disease which limits exercise and COPD and blood pressure is not controlled;
2. not suffering serious vision problems;
3. does not suffer from this problem: (a score of 24 or higher on MOCA);
4. a year after analyzing the type of hip replacement or knee or broken extremities;
5. Does not suffer any neurological diseases or stroke.

Ages: 70 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The step recovery thresholds and brain imaging (MRI) | 60 minute
  The stepping threshold as measured by the distance of the platform movements in centimeters will be measured. Quantitative parameters of the compensatory stepping/ and motor ability (i.e., step reaction time, step time, step length), descriptive parameters of the stepping strategy after perturbation (i.e., arm responses, upper body responses, leg step threshold and fall threshold). In addition we will be testing the correlation between brain activity using brain imaging in both to find whether improvement in motor function are correlated with brain function and anatomy.

SECONDARY OUTCOMES:
Postural stability | 10 minutes
  participants will be instructed to stand upright on the force platform with the feet positioned as close as possible (heels and toes touching). A total of six 30-second trials will conduct for two visual conditions: eyes open and eyes closed. Balance measurements will be collected with a Kistler 9287 single force platform (Kistler Instrument Corp, Winterthur, Switzerland), which measures the time-varying displacement of the center of pressure (CoP) under the participant's feet. The force platform data will be sampled at a frequency of 100 Hz and stored on a hard disk for later processing.
Voluntary step test | 6 minutes
  subjects will be instructed to step as quickly as possible following a cue signal
Berg Balance test | 10 minutes
  The participant is scored on 14 balance tasks. Maximum score of 56 represents good balance. Higher scores indicate higher levels of balance function, while 45 or less indicates a high risk of falling.
kinematics of walking | 10 minutes
  subjects will be instructed to walk on a treadmill. During the experiment we will measure by 3D motion analysis system gait kinematics during walking at their preferred speed for 2 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: ilan Shelef, MD, Study Chair — Soroka University Medical Center
Locations (3):
- Israel (3):
  - Ben-guion University of the Negev,, Beersheba
  - Soroka Medical Center, Beersheba
  - SorokaUMC, Beersheba

REFERENCES:
- [Derived] Paran I, Nachmani H, Salti M, Shelef I, Melzer I. Balance recovery stepping responses during walking were not affected by a concurrent cognitive task among older adults. BMC Geriatr. 2022 Apr 6;22(1):289. doi: 10.1186/s12877-022-02969-w. PMID 35387589
- [Derived] Nachmani H, Paran I, Salti M, Shelef I, Melzer I. Examining Different Motor Learning Paradigms for Improving Balance Recovery Abilities Among Older Adults, Random vs. Block Training-Study Protocol of a Randomized Non-inferiority Controlled Trial. Front Hum Neurosci. 2021 Feb 25;15:624492. doi: 10.3389/fnhum.2021.624492. eCollection 2021. PMID 33716695